CLINICAL TRIAL: NCT02399423
Title: The GlasVEGAS Study (Glasgow Visceral & Ectopic Fat With Weight Gain in South AsianS) - Does Adipose Tissue Expandibility Differ Between South Asians and Europeans and Does This Contribute to Differences in Cardio-metabolic Disease Risk?
Brief Title: The GlasVEGAS Study (Glasgow Visceral & Ectopic Fat With Weight Gain in South AsianS)
Acronym: GlasVEGAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Göteborg University (Other); University of Pisa (Other)
Responsible Party: Principal Investigator, Professor Naveed Sattar, Professor of Metabolic medicine, University of Glasgow
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Project number 60315/1
Record Dates: First submitted 2015-03-12; First posted 2015-03-26 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Diabetes; Weight Gain; Weight Loss; Cardiovascular Disease; Obesity
Keywords: diabetes; metabolism; cardiovascular disease; weight gain; weight loss; european; south asian; obesity
MeSH Terms: conditions — Diabetes Mellitus; Weight Gain; Weight Loss; Cardiovascular Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- South Asian participants (Other): 30 South Asian male participants
  Interventions: Behavioral: Weight gain; Behavioral: Weight loss
- European participants (Other): 30 European male participants
  Interventions: Behavioral: Weight gain; Behavioral: Weight loss

INTERVENTIONS:
Behavioral: Weight gain — Weight gain of 7% body weight over 4-6 weeks by ingesting an extra 1500-2000 kcal/day
Behavioral: Weight loss — Weight loss of 7-15% body weight over 12 weeks by increased exercise and either an alternate day fasting dietary regime or a weight watchers dietary regime

SUMMARY:
South Asians have a much higher risk of diabetes compared to Europeans and investigators don't know why this is. Investigators think that South Asians' capacity to store fat safely under the skin is lower than Europeans, so they start to store fat around internal organs and in liver and muscle, and at lower body weights than Europeans. These increased levels of internal fat storage are thought to increase risk of diabetes.

The purpose of the study therefore is to investigate whether there are differences with weight gain and weight loss in fat storage, fat cell function and metabolic risk factors, in South Asians compared with Europeans. Investigators will compare South Asian and European men at the start of the study, after they have gained about 7% body weight, and again after they have lost 7-15% body weight (from peak weight) to see how gaining and losing weight affects fat storage within the body and the function of fat cells. Investigators will also assess the effect of weight gain and weight loss on metabolism, fitness and risk factors for diabetes and heart disease.

DETAILED DESCRIPTION:
South Asians have about five times the risk of adult onset diabetes (high blood sugar) than Europeans and nearly one in five South Asian men in the United Kingdom have the disease. Diabetes is a serious disease that can lead to a number of adverse health consequences including heart disease, kidney disease and blindness and accounts for about 10% of all healthcare costs in the UK. Obesity is strongly linked to diabetes risk, but the adverse effect of getting fatter on diabetes risk is much higher in South Asians than Europeans. The purpose of this study is to understand why this is the case. When humans put on weight initially this fat is stored under the skin (subcutaneous fat). This is relatively safe. However, when the capacity of this under skin storage is exceeded, fat is stored internally within the tummy area (visceral fat) and in organs such as the liver and muscle, which is less safe and increases diabetes risk. Investigators think that South Asians' capacity to store fat safely under the skin is lower than Europeans, so fat is stored internally and in liver and muscle at lower body weights than Europeans. The purpose of this study is to investigate whether this occurs and why. To do this investigators will compare a group of South Asian and European men and see how gaining and losing weight affects fat storage within the body and the function of fat cells. Investigators will also assess the effect of weight gain and weight loss on metabolism, fitness and risk factors for diabetes and heart disease.

The study will include healthy men of normal weight aged between 18-45 year and of either white European or South Asian (both parent of Indian, Pakistani, Bangladesh or Sri Lankan origin) ethnic origin.

Body weight will be altered by initially gaining weight and then losing weight. To do this participants will initially have to eat more food for 4-6 weeks and then go on a diet combined with exercise for 12 weeks. Participation in the study will last around 5½ months in total.

During the study pictures of body fat stores will be taken using an MRI scanner, a biopsy/sample of tummy fat will be taken to look at the fat cells and physical fitness and body metabolism (the way the body deals with sugar, insulin and fat) will be measured. These measurements will be done at three different times: before gaining weight, once weight is gained, and after losing weight (and back to original weight). The measurements will give a detailed assessment of the changes in the body when gaining or losing weight.

The benefits of taking part in the study are receiving detailed feedback about fitness levels, body fat, dietary intake, blood pressure, cholesterol, blood sugar and level of "insulin resistance". Feedback about the overall study findings will also be provided.

In addition, the knowledge gained from participation may benefit people who are at risk of diabetes in the future by increasing our understanding of why South Asians are at increased risk of developing diabetes. It will also help guide future research investigating how to reduce this increased risk through lifestyle changes and may also help direct the development of medicines to prevent and treat diabetes groups at increased risk of the disease.

Possible disadvantages of the study are gaining 7% of body weight over 4-6 weeks. This is likely to temporarily induce negative metabolic changes. However, investigators are also supporting losing this weight (and hopefully more) in the weight loss phase of the study. There is no evidence that short-term weight gain of this nature causes any long-term adverse effects. Longer-term weight gain however is associated with an increased risk of diabetes, cardiovascular disease and high blood pressure. It is therefore important that investigators ensure participants return to original weight at the start of the study. Taking fat biopsies carries a small risk of minor bruising or an infection. Good sterile practice reduces this risk of infection and application of ice and pressure to the biopsy site reduces the risk of bruising. Blood sampling via the cannula may cause minor bruising or an inflammation of the vein. Some participants may feel faint when they give blood. One of the exercise tests will be at a maximal level and the possibility exists that, very occasionally, certain changes may occur during or shortly after the test. They include abnormal blood pressure, fainting or a change in the normal rhythm of the heartbeat. There is a small possibility that taking part in this study will reveal a health problem that patients already have such as high cholesterol or high blood pressure. If such a problem is revealed, investigators will ask permission to inform the participant's General Practitioner to receive clinically appropriate follow-up care.

This study is running for ~2.5 years from March 2015 and is based at the University of Glasgow. The study is being funded by the European Commission as part of the European Medical Information Framework (EMIF), called EMIF-Metabolic. This research will help investigators to better predict who is likely to be at risk of developing diseases such as diabetes and to develop new medicines to prevent and treat these diseases. More details about EMIF-Metabolic are available here: http://www.emif.eu/emif-meta/objectives.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be men of European (self-report of both parents of white European origin) or South Asian (self-report of both parents of Indian, Pakistani, Bangladeshi or Sri Lankan origin) with BMI <25 kg.m-2, who have been weight stable (± 2 kg) for >6 months.

Exclusion Criteria:

* Exclusion criteria will include diabetes (physician diagnosed or HbA1c ≥6.5% on screening), history of cardiovascular disease, regular participation in vigorous physical activity, current smoking, taking drugs or supplements thought to affect carbohydrate or lipid metabolism, or other significant illness that would prevent full participation in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Change in body metabolism after gaining 7% body weight and after losing 7% of body weight | Weight gain assessment made after an expected average of 5 weeks and weight loss assessment after 12 weeks
  Metabolic changes will be calculated by measuring levels of insulin, c-peptide, glucose, non-esterified fatty acids and NMR metabolomic responses to a standard 800 kcal meal tolerance test over 5 hours. Fasting serum adipokine levels will also be taken. Metabolic rate and substrate utilisation will be measured by indirect calorimetry using a ventilated hood.
Change in visceral adipose tissue after gaining 7% body weight and after losing 7% body weight | Weight gain assessment made after an expected average of 5 weeks and weight loss assessment after 12 weeks
  Adipose tissue will be measured by MRI scanner and the change in visceral adipose tissue quantified
Change in subcutaneous adipose tissue after gaining 7% body weight and after losing 7% body weight | Weight gain assessment made after an expected average of 5 weeks and Weight loss assessment after 12 weeks
  Adipose tissue will be measured by MRI scanner and the change in subcutaneous adipose tissue quantified.
Change in liver adipose tissue after gaining 7% body weight and after losing 7% body weight | Weight gain assessment made after an expected average of 5 weeks and Weight loss assessment after 12 weeks
  Liver adipose tissue will be measured by MRI spectroscopy and the change in liver adipose tissue quantified.
Change in adipose cell morphology after gaining 7% body weight and after losing 7% body weight. | Weight gain assessment made after an expected average of 5 weeks and weight loss assessment after 12 weeks
  Adipose cells will be obtained by needle biopsy from the subcutaneous layers of adipose tissue in the abdomen. Following this adipose cells will be assessed for their morphology including size and number.
Change in adipose cell insulin sensitivity after gaining 7% body weight and after losing 7% body weight | Weight gain assessment made after an expected average of 5 weeks and weight loss assessment after 12 weeks
  Adipose cells will be obtained by needle biopsy from the subcutaneous layers of adipose tissue in the abdomen. Following this adipose cells will be assessed for their sensitivity to insulin.
Change in adipose cell function after gaining 7% body weight and after losing 7% body weight | Weight gain assessment made after an expected average of 5 weeks and weight loss assessment after 12 weeks
  Adipose cells will be obtained by needle biopsy from the subcutaneous layers of adipose tissue in the abdomen. Following this adipose cells will be assessed for their cell function including gene expression markers related to triglyceride storage and differentiation of the cells.

SECONDARY OUTCOMES:
Change in fitness after gaining 7% body weight and after losing 7% of body weight | Weight gain assessment made after an expected average of 5 weeks and weight loss assessment after 12 weeks
  Fitness will be assessed by an incremental uphill treadmill walking protocol. Maximal oxygen uptake (VO2) max will then be calculated as a measure of fitness.
Change in physical activity after gaining 7% body weight and after losing 7% of body weight | Weight gain assessment made after an expected average of 5 weeks and weight loss assessment after 12 weeks
  Physical activity will be measured objectively by accelerometer
Change in dietary intake after gaining 7% body weight and after losing 7% of body weight | Weight gain assessment made after an expected average of 5 weeks and weight loss assessment after 12 weeks
  Dietary intake will be measured by weighed food record
Change in facial appearance after gaining 7% body weight and after losing 7% of body weight | Weight gain assessment made after an expected average of 5 weeks and weight loss assessment after 12 weeks
  An additional optional component of the study is to have digital photographs taken which has been shown to correlate to health status. The photographs will be assessed by computer and analysed anonymously.
Change in qualitative interviews after gaining 7% body weight and after losing 7% of body weight | Weight gain assessment made after an expected average of 5 weeks and weight loss assessment after 12 weeks
  An additional optional component of the study is qualitative interviews to assess body image, self-esteem and psychological wellbeing during the study.
Change in cognition after gaining 7% body weight and after losing 7% of body weight | Weight gain assessment made after an expected average of 5 weeks and weight loss assessment after 12 weeks
  An additional option as part of the study is to assess cognition by means of a Sensitive Cognitive Assessment Inventory (SCAI) assessment tool. This involves a computer test which will assesses indices of cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Sattar, MD PhD, Principal Investigator — Univesity of Glasgow; Jason MR Gill, PhD, Principal Investigator — Univesity of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

REFERENCES:
- [Derived] Beazer JD, McLaren J, Christoffersen C, Ferraz MJ, Mulder MT, Graham D, Karlsson H, Ljunggren SA, Gill JMR, Freeman DJ. HDL protein composition differs between young white European and South Asian men before and after weight gain. Clin Sci (Lond). 2025 Dec 18;139(24):1659-74. doi: 10.1042/CS20258040. PMID 41416660
- [Derived] McLaren J, Gao X, Ghouri N, Freeman DJ, Richardson J, Sattar N, Gill JMR. Weight gain leads to greater adverse metabolic responses in South Asian compared with white European men: the GlasVEGAS study. Nat Metab. 2024 Aug;6(8):1632-1645. doi: 10.1038/s42255-024-01101-z. Epub 2024 Aug 16. PMID 39152223